CLINICAL TRIAL: NCT05545709
Title: Clinical Application of 5G-based Telerobot-assisted Spine Surgery
Brief Title: 5G-based Telerobot-assisted Spine Surgery
Status: Completed | Type: Observational
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Wei Tian, Clinical Professor, Beijing Jishuitan Hospital
Other Study IDs: JST 202005-08
Record Dates: First submitted 2022-09-12; First posted 2022-09-19 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- remote group: Based on the 5G network, the orthopedic robotic remote surgery platform is built at Beijing Jishuitan Hospital, providing primary hospitals with a platform for preoperative consultation, intraoperative communication and surgical robot teleoperation, and postoperative follow-up. With the support of the 5G network, equipment and surgical robots are integrated into the remote surgery service platform, building a high-speed transmission channel between Beijing Jishuitan Hospital and other hospitals.
  Interventions: Procedure: remote robot-assisted spine surgery
- local group: Local orthopedic robot-assisted spine surgeries were performed according to the guidelines for thoracolumbar pedicle screw placement assisted by orthopedic surgical robots.

INTERVENTIONS:
Procedure: remote robot-assisted spine surgery — Based on the 5G network, the orthopedic robotic remote surgery platform is built at Beijing Jishuitan Hospital, providing primary hospitals with a platform for preoperative consultation, intraoperative communication and surgical robot teleoperation, and postoperative follow-up. With the support of the 5G network, equipment and surgical robots are integrated into the remote surgery service platform, building a high-speed transmission channel between Beijing Jishuitan Hospital and other hospitals.
  Groups: remote group

SUMMARY:
This study retrospectively analyzed cases of remote robot-assisted spine surgery performed jointly by the Beijing Jishuitan Hospital Spinal Surgery and partner hospitals, with cases of local orthopedic robot-assisted spine surgeries performed by Beijing Jishuitan Hospital between April 2021 and December 2021.

DETAILED DESCRIPTION:
Local orthopedic robot-assisted spine surgeries were performed according to the guidelines for thoracolumbar pedicle screw placement assisted by orthopedic surgical robots.

Based on the 5G network, the orthopedic robotic remote surgery platform is built at Beijing Jishuitan Hospital, providing primary hospitals with a platform for preoperative consultation, intraoperative communication and surgical robot teleoperation, and postoperative follow-up. With the support of the 5G network, equipment and surgical robots are integrated into the remote surgery service platform, building a high-speed transmission channel between Beijing Jishuitan Hospital and other hospitals.

ELIGIBILITY:
Inclusion Criteria:

* patients received remote robot-assisted spinal surgery or local orthopedic robot-assisted spinal surgery;
* patients had complete medical records and imaging data;
* patients provided informed consent.

Exclusion Criteria:

* revision surgery;
* more than four surgical segments;
* patients with severe comorbidities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients accepted robot-assisted spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The accuracy of guide-wire placement or positioning | 1 month
  according to the Gertzbein and Robbins scale, including grade A (screw was completely within the pedicle), grade B (pedicle cortical breach <2 mm), grade C (pedicle cortical breach <4 mm), grade D (pedicle cortical breach <6 mm), and grade E (pedicle cortical breach >6 mm).

SECONDARY OUTCOMES:
operation time | 1 day
  Time from start to finish of surgery
complication | 1 month
  Nerve injury, epidural hematoma, and infection
network interruptions | 1 day
  failure to establish connection, the interruption of connection and severe delays in connection, and remote surgery abandonment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No